CLINICAL TRIAL: NCT04961697
Title: Family and Patient Outcomes After Pediatric Intensive Care
Brief Title: Family and Patient Outcomes After Pediatric Intensive Care (FOREVER)
Acronym: FOREVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: FOREVER
Record Dates: First submitted 2021-06-22; First posted 2021-07-14 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Post-Intensive Care Syndrome; Anxiety; Depression; Stress Disorders, Post-Traumatic; Quality of Life; Satisfaction, Patient
Keywords: Post-Intensive Care Syndrome; Anxiety; Depression; Post-Traumatic Stress Disorder; Health-related Quality of Life; Satisfaction with Care
MeSH Terms: conditions — postintensive care syndrome; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This is a multicentric two-arm two-period crossover study: in the first phase each PICU will be randomized between intervention (PICU with diaries) and control (PICU without diaries), crossing over in the second phase after a washout period.
Who Masked: Outcomes Assessor
Masking Description: Since the intervention is the use of hospital diaries there will be masking in the outpatient follow-up data collection and posterior data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICU with diaries (Experimental): The main family member of a critically ill child will receive a diary upon PICU admission.
  Except for the diaries intervention, this group of patients will be submitted to usual PICU routine care.
  Interventions: Behavioral: Hospital diaries
- PICU without diaries (No Intervention): This group of critically ill patients and family members will not receive diaries, but will also be submitted to usual PICU routine care.

INTERVENTIONS:
Behavioral: Hospital diaries — Diaries will be used by family members, PICU staff or even the patient himself. They will take daily notes expressing feelings and thoughts and describing events that might help chronologically to better understand the course of disease and PICU stay. Photographs and other important PICU memories may also be used in the diary.
  Arms: PICU with diaries

SUMMARY:
This study aims to evaluate in the Brazilian context, the impact of the implementation of a diary program on patient and family-centered outcomes after PICU discharge. The intervention investigated will be the use of hospital diaries for the critically ill child in a cross-over study, randomized by clusters in four PICUs of Rio de Janeiro. Family members of children aged 29 days to 12 years, admitted for more than 36 hours will be included and data collection will take place upon admission, at PICU discharge and 60 days after discharge from the PICU.

Family-centered outcomes assessed will be: satisfaction with care, anxiety and depression at discharge, incidence of anxiety, depression, PTSD, burden and quality of life in follow-up. Patient-centered outcomes will be assessed in children at discharge and follow-up - quality of life and incidence of new morbidities will be evaluated. The association of clinical, social and demographic variables with family- and patient-centered outcomes will be investigated on an exploratory basis. Burnout Syndrome in PICU health professionals will be assessed before and after the intervention as a proxy of intervention security for PICU staff.

DETAILED DESCRIPTION:
More than one third of parents and patients admitted to Pediatric Intensive Care Units (PICU) develop Anxiety, Depression and Posttraumatic Stress Disorder (PTSD), with consequent decrease in quality of life and great social impact, known as Pediatric and Family Post-Intensive Care Syndrome (PICS and PICS-F). Strategies that minimize negative outcomes after discharge have been adopted, such as the use of hospital diaries to regularly record the impressions of family members and health professionals about the patient's evolution, hosting parents and encouraging their direct participation in care.

This study aims to evaluate in the Brazilian context, the impact of the implementation of a diary program on patient and family-centered outcomes after discharge. The intervention investigated will be the use of hospital diaries for the critically ill child in a cross-over study, randomized by clusters in four PICUs of Rio de Janeiro, totaling 200 family members in the intervention group and 200 controls. Family members of children aged 29 days to 12 years, admitted for more than 36 hours will be included and data collection will take place upon admission, at discharge and 60 days after discharge from the PICU. Family-centered outcomes assessed will be: satisfaction with care, anxiety and depression at discharge, incidence of anxiety, depression, PTSD, burden and quality of life in follow-up. Quality of life and incidence of new morbidities will be evaluated in children at discharge and follow-up, as well as Burnout Syndrome in the health team. The association of clinical, social and demographic variables with family- and patient-centered outcomes will be investigated on an exploratory basis.

With this study, we aim to contribute to a better knowledge about different family-centered outcomes in intensive care, allowing reduction of health problems and the development of policies that seek to alleviate suffering, to humanize intensive environments and encourage participation of family members in child care during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients between age limits admitted in PICU for clinical or surgical reasons with 36 or more hours of stay and their main family member.
* Physicians, registered nurses, nurse technicians, physical therapists and other professionals working in participants PICU involved in caring for patients and their families and taking notes in the diaries

Exclusion Criteria:

* Patients admitted for monitorization or elective low-complexity surgeries
* Patients readmitted between the first admission and the first follow-up visit
* Patients in palliative care
* Families with linguistic or comprehension barriers
* Families residencies situated outside Rio de Janeiro metropolitan region

Ages: 29 Days to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 431 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Incidence of anxiety symptoms in family member from critically ill child. | 45-60 days after PICU discharge
  Proportion of main family member positive for anxiety symptoms as measured by HADS (Hospital Anxiety and Depression Scale from Zigmond and Snaith), a self-report standardized 14-item questionnaire covering an anxiety 7-question subscale and a depression 7-question subscale. Each subscale includes Likert-scaled questions ranging from 0 to 3. Presence of anxiety symptoms will be determined when 9 or more points on each subscale.
Incidence of depression symptoms in family member from critically ill child. | 45-60 days after PICU discharge
  Proportion of main family member positive for depression symptoms as measured by HADS (Hospital Anxiety and Depression Scale from Zigmond and Snaith), a self-report standardized 14-item questionnaire covering an anxiety 7-question subscale and a depression 7-question subscale. Each subscale includes Likert-scaled questions ranging from 0 to 3. Presence of depression symptoms will be determined when 9 or more points on each subscale.
Incidence of PTSD (Posttraumatic Stress Disorder) in family member from critically ill child. | 45-60 days after PICU discharge
  Proportion of main family member positive for PTSD as measured by PCL-5 (Posttraumatic Stress Disorder Checklist for DSM-V - Diagnostic and Statistical Manual of Mental Disorders - V from Weathers et al), a self-report standardized 20-item questionnaire covering four dimensions of symptoms: intrusions, avoidance, negative alterations in cognitions and mood and alterations in arousal and reactivity. Each subscale includes Likert-scaled questions ranging from 0 (not at all) to 4 (extremely). Presence of PTSD symptoms when 33 or more total points or positivity in each DSM-V dimension.

SECONDARY OUTCOMES:
Evaluate family satisfaction with PICU care as measured by EMpowerment of PArents in THe Intensive Care 30 (EMPATHIC-30) questionnaire. | Until 72 hours after the patient discharge from Pediatric Intensive Care Unit
  Quantify family satisfaction with PICU care as measured by EMPATHIC-30 (Latour et al), a self-report standardized 30-item questionnaire covering 5 domains: information, care and treatment, organization, parent participation and professional attitude. Each subscale includes Likert-scaled questions ranging from 1 (certainly no) to 6 (certainly yes). Higher scores, higher family satisfaction with care.
Evaluate alterations in family quality of life as measured by Short Form 12 (SF-12) questionnaire | 45-60 days after PICU discharge
  Quantify family quality of life as measured by SF-12 (Ware et al), a self-report standardized 12-item questionnaire covering a mental and a physical component, with Likert-scaled questions ranging variedly. Higher scores, better quality of life.
Incidence of Anxiety and Depression in family members of a critically ill child using HADS instrument upon PICU discharge. | Until 72 hours after the patient discharge from Pediatric Intensive Care Unit
  Proportion of main family member positive for anxiety and depression as measured by HADS (Zigmond and Snaith), a self-report standardized 14-item questionnaire covering an anxiety 7-question subscale and a depression 7-question subscale. Each subscale includes Likert-scaled questions ranging from 0 to 3. Presence of anxiety or depression symptoms when 9 or more points on each subscale.
Incidence of New Morbidity in critically ill children at PICU discharge. | Until 72 hours after the patient discharge from Pediatric Intensive Care Unit
  Incidence of New Morbidities in critically ill children admitted to a PICU, measured using the Functional Status Scale (FSS) upon admission, at PICU discharge and 60 days after PICU discharge. A raise in 3-points in FSS total score will be described as "New Morbidity", as assigned by Pollack et al.
Incidence of New Morbidity in critically ill children after PICU discharge. | 45-60 days after PICU discharge
  Incidence of New Morbidities in critically ill children admitted to a PICU, measured using the Functional Status Scale (FSS) upon admission, at PICU discharge and 60 days after PICU discharge. A raise in 3-points in FSS total score will be described as "New Morbidity", as assigned by Pollack et al.
Evaluate alterations in critically ill children Quality of Life as measured by Pediatric Quality of Life Questionnaire (PedsQL). | 45-60 days after PICU discharge
  Quantify critically ill children Quality of Life after PICU discharge as measured by Pediatric Quality of Life Questionnaire (PedsQL).
Prevalence of Burden in the main family member after PICU discharge measured with Zarit Burden Scale. | 45-60 days after PICU discharge
  Prevalence of Burden in the main family member of a critically ill child after PICU discharge measured with Zarit Burden Scale (ZBI). This scale consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. Higher scores indicate greater burden.
Perceptions of health professionals regarding the use of PICU diaries | One-month after the intervention period, which ends after the inclusion of 50 patient's family-members.
  Perceptions of health professionals regarding the use of PICU diaries using a semi-structured questionnaire specifically developed for this study
Perceptions of parents and main family members of a critically ill child regarding the use of PICU diaries | 45-60 days after PICU discharge upon intervention period
  Perceptions of parents and main family members of a critically ill child regarding the use of PICU diaries using a semi-structured questionnaire specifically developed for this study
Evaluate alterations in the three dimensions of the Maslach Burnout Inventory - emotional exhaustion, depersonalization and personal accomplishment - in PICU health professional. | One month before the beginning of the intervention in the PICU and one-month after the end of intervention period, which ends after the inclusion of 50 patient's family-members.
  Evaluate alterations in PICU staff Burnout Syndrome scores, measured in the three dimensions of the Maslach Burnout Inventory - emotional exhaustion, depersonalization and personal accomplishment, as a proxy of intervention security for health professionals.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Lima-Setta, Principal Investigator — D'Or Institute for Research and Education
Locations (1):
- D'Or Institute for Research and Education, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Harvey MA. The truth about consequences--post-intensive care syndrome in intensive care unit survivors and their families. Crit Care Med. 2012 Aug;40(8):2506-7. doi: 10.1097/CCM.0b013e318258e943. No abstract available. PMID 22809925
- [Background] Huggins EL, Bloom SL, Stollings JL, Camp M, Sevin CM, Jackson JC. A Clinic Model: Post-Intensive Care Syndrome and Post-Intensive Care Syndrome-Family. AACN Adv Crit Care. 2016 Apr-Jun;27(2):204-11. doi: 10.4037/aacnacc2016611. PMID 27153309
- [Background] Myers EA, Smith DA, Allen SR, Kaplan LJ. Post-ICU syndrome: Rescuing the undiagnosed. JAAPA. 2016 Apr;29(4):34-7. doi: 10.1097/01.JAA.0000481401.21841.32. PMID 27023654
- [Background] Svenningsen H, Langhorn L, Agard AS, Dreyer P. Post-ICU symptoms, consequences, and follow-up: an integrative review. Nurs Crit Care. 2017 Jul;22(4):212-220. doi: 10.1111/nicc.12165. Epub 2015 Feb 17. PMID 25688675
- [Background] Davidson JE, Aslakson RA, Long AC, Puntillo KA, Kross EK, Hart J, Cox CE, Wunsch H, Wickline MA, Nunnally ME, Netzer G, Kentish-Barnes N, Sprung CL, Hartog CS, Coombs M, Gerritsen RT, Hopkins RO, Franck LS, Skrobik Y, Kon AA, Scruth EA, Harvey MA, Lewis-Newby M, White DB, Swoboda SM, Cooke CR, Levy MM, Azoulay E, Curtis JR. Guidelines for Family-Centered Care in the Neonatal, Pediatric, and Adult ICU. Crit Care Med. 2017 Jan;45(1):103-128. doi: 10.1097/CCM.0000000000002169. PMID 27984278
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] Elliott D, Davidson JE, Harvey MA, Bemis-Dougherty A, Hopkins RO, Iwashyna TJ, Wagner J, Weinert C, Wunsch H, Bienvenu OJ, Black G, Brady S, Brodsky MB, Deutschman C, Doepp D, Flatley C, Fosnight S, Gittler M, Gomez BT, Hyzy R, Louis D, Mandel R, Maxwell C, Muldoon SR, Perme CS, Reilly C, Robinson MR, Rubin E, Schmidt DM, Schuller J, Scruth E, Siegal E, Spill GR, Sprenger S, Straumanis JP, Sutton P, Swoboda SM, Twaddle ML, Needham DM. Exploring the scope of post-intensive care syndrome therapy and care: engagement of non-critical care providers and survivors in a second stakeholders meeting. Crit Care Med. 2014 Dec;42(12):2518-26. doi: 10.1097/CCM.0000000000000525. PMID 25083984
- [Background] Jezierska N. Psychological reactions in family members of patients hospitalised in intensive care units. Anaesthesiol Intensive Ther. 2014 Jan-Mar;46(1):42-5. doi: 10.5603/AIT.2014.0009. PMID 24643927
- [Background] Davidson JE, Jones C, Bienvenu OJ. Family response to critical illness: postintensive care syndrome-family. Crit Care Med. 2012 Feb;40(2):618-24. doi: 10.1097/CCM.0b013e318236ebf9. PMID 22080636
- [Background] Goldfarb MJ, Bibas L, Bartlett V, Jones H, Khan N. Outcomes of Patient- and Family-Centered Care Interventions in the ICU: A Systematic Review and Meta-Analysis. Crit Care Med. 2017 Oct;45(10):1751-1761. doi: 10.1097/CCM.0000000000002624. PMID 28749855